CLINICAL TRIAL: NCT02200068
Title: Usual Care Randomized Study Measuring the Impact of an Online Personal Health Record (Sanoia) in Rheumatoid Arthritis Patients on Reported Outcomes
Brief Title: CARNet : Self-Monitoring and Co-driving in Rheumatology With Internet : Rheumatoid Arthritis Cohort (Usual Care Study)
Acronym: CARNet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Accompagnement pour un Internet en Médecine et Santé au Service des Usagers (Other)
Collaborators: UCB France S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2013-A00105-40
Record Dates: First submitted 2014-07-09; First posted 2014-07-25 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Perceived Efficacy of Patient Physician Interactions; Patient Reported Outcomes; Personal Health Record
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PHR Group (Active Comparator): This group will have access to a personal health record website SANOIA in addition to all resources they use or find online
  Interventions: Other: SANOIA Website
- Non-PHR Group (No Intervention): This group will not be informed of the Personal Health Record Website and will use Internet as they usually do.

INTERVENTIONS:
Other: SANOIA Website
  Arms: PHR Group

SUMMARY:
Recommendations of Rheumatoid Arthritis management agree on the necessity of patient self-involvement in the care. In parallel, the observation of the adoption rate of websites directed toward patients may indicate that this involvement is shared by a large number ot the population.

However, most of these sites are only informative and few of them offer patients to be engaged to generate their own data that can impact on the patient-physician relationship by easing the dialog and then leading to better mutual understanding.

As new web or mobile services allowing patients to self-report their outcomes are flourishing only a very few of them have already addressed the their impact of the patient-physician relationship.

The main objective of this study is to quantify the effect of a website (Sanoia) on the quality of patient-doctor interactions, as perceived by the patient using the french translations of the Peppi Questionnaire during the 12 months observation period.

In France, the patient protection committee (CPP) has ranked this study in "Soins Courants" (Usual Care).

DETAILED DESCRIPTION:
Recommendations of care in rheumatoid arthritis (RA) advocate for patient involvement and management of his/her own health.

The observation of the sole rate of use of websites specialized health patients might indicate that this involvement is occurring for a large number. Indeed, yet in 2010, more than 71% of French Netizen used the Internet to search for information related to their health according to a 2012 survey from the French National Order of Medical Doctors. Focusing on rheumatology, 68% of French patients have already used the Internet to search for information related to their arthritis as shown from a 2012 survey of the French Society of Rheumatology. In this medical field, these results reflect the fact that in France since years 2000, patients' associations and institutions, edited websites to offer patients a direct and easier access to information on diseases or treatments.

Nevertheless, it is useful to observe the type of service provided to the patient on these sites: the majority of these sites, even the most recent offer only the dissemination of information and never have been studied on this informative nature. These sites should be considered as an introductory step toward patient involvement.

Indeed, patients involvement is effective if they are really "active" and produce data, e.g. when him(her)self notes personal information online, manages a 'health book' virtual or self-assessing internet. In other words, involvement makes sense when it contributes to an "improvement" doctor-patient exchanges and when at last it leads to an increase in entropy.

Especially the latter type of use, i.e. the patient self-reported measure (patient-reported outcomes), can be a manner to both involve the patient in his care, and to feed the medical decision support with the certified rheumatologist. Moreover, it appears that the self-measurements in particular by the RA patient, are reliable.

In recent years, new services on the web or mobile begun to address this need and allowed patients to report issues relating to their health (current treatments, etc..), and to perform self-measures (pain, activity, morning stiffness, etc..). Notwithstanding visibility increasingly strong, it is striking to note that these tools, including those for self-measurement, have been little evaluated in terms of impact, for example on doctor-patient exchanges.

Indeed, Investigators have chosen to measure the characteristics of these exchanges, as perceived by the patient: effectiveness, quality and overall quality of care using dedicated tools.

In France, the patient protection committee (CPP) has ranked this study in "Soins Courants" (Usual Care).

The study will use the web-based platform (*) Sanoia.com, partner of the French Society of Rheumatology, which provides a trusted environment to its users via anonymity. This platform is recognized as innovative by the French Ministry of Research and relies on a data hosting architecture approved by the Ministry of Health. The statistical analysis of users data is limited to research purposes and placed under the dual supervision of patient associations and medical societies. These features are the source of its success in terms of audience with patients (> 145,000 health records created in September 2012).

Specifically Sanoia offers, among other benefits, Rheumatoid Arthritis (RA) patients to list their medical history and access to tools for self-measures, whether generic (e.g. notepad symptoms, followed by medications taken, etc.), or more specific to RA (e.g. RAPID3: routine assessment of patient index data, Health Assessment Questionnaire, Rheumatoid Arthritis Impact of Disease (RAID) score. Based on these data, a customized selection of information (based on an Internet monitoring performed by patient association ANDAR and validated by the medical society SFR) is displayed.

The main objective of this study is to quantify with RA patients the effect of a website (Sanoia) on the quality of patient-doctor interactions, as perceived by the patient using the french translations of the physician investigator to investigate the perceived efficacy ot the patient-physician relationship (PEPPI) Questionnaire during the 12 months observation period.

(*) : SANOIA is a personal health record platform that does not embed or to connect to social networks.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 years.
* Patient with Rheumatoid Arthritis diagnosed according to American College of Rheumatology (ACR ) / European League Against Rheumatism (EULAR) 2010 criteria.
* Patient monitored by the recruiting physician from over a year.
* Patient access who have access to an Internet broadband equipment other than on a mobile or a a smartphone

Exclusion Criteria:

* Patient already using Sanoia at the time of inclusion.
* Patient already participating in a therapeutic clinical trial in rheumatology
* Patient having no computer literacy and understanding difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 12 months after inclusion of Perceived efficacy by the patient of patient-physician interactions (PEPPI) | Baseline and Month 12
  Patients connects to the electronic Case Report Form (e-CRF) and file the French translation of the 5-item PEPPI Questionnaire

SECONDARY OUTCOMES:
Rheumatoid Arthritis Impact of Disease (RAID) score | Baseline, Month 3, Month 6 and Month 12
  Patients connects to the e-CRF and file the French translation of the Rheumatoid Arthritis Impact of Disease (RAID) score
Overall assessment of the patient's Health as measured by a VAS | Baseline, Month 3, Month 6 and Month 12
  Patients connects to the e-CRF and move a cursor on the appropriate value on a Visual Analogic Scale
Patient-Physician communication quality, as assessed by the patient using a Numeric Rating Scale | Baseline, Month 3, Month 6 and Month 12
  Patients connects to the e-CRF and selects the appropriate number on a Numeric Rating scale
Overall perceived quality of care, as assessed by the patient via a Numeric Rating Scale | Baseline, Month 3, Month 6 and Month 12
  Patients connects to the e-CRF and selects the appropriate number on a Numeric Rating scale
Number of patient's visits to the Rheumatologist from baseline to 12 months after inclusion | Month 3, Month 6 and Month 12
  Patient reports the number of visits to the Rheumatologist
Satisfaction of SANOIA using a Numeric Rating Scale for the PHR Group | Month 3 and Month 12
  Patients connects to the e-CRF and selects the appropriate number on a Numeric Rating scale
Unsatisfactory criteria using a pre-defined list for the PHR Group | Month 3 and Month 12
  Patients connects to the e-CRF and selects the appropriate items in a list of pre-defined criteria
Spontaneous access and use of SANOIA for Non-PHR Group (usual care) | Month 12
  Time period and origin of access of Group 2 Patients (usual care) that incidentally used SANOIA prior or during the study
Health Assessment Quality of Life Disability Index Questionnaire | Baseline
  Patients connects to the e-CRF and file the French translation of the Health Assessment Quality of Life Disability Index Questionnaire
Co-morbidities list | Baseline
  Patients connects to the e-CRF and file the French translation of the 15 item (12 compulsory answers and 3 additional open items) of an adapted Comorbidities Questionnaire

OTHER OUTCOMES:
Value of Perceived efficacy by the patient of patient-physician interactions (PEPPI) | Month 3 and Month 6
  Patients connects to the electronic Case Report Form (e-CRF) and file the French translation of the 5-item PEPPI Questionnaire

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - University Hospital Jean Minjoz, Besançon
  - Chu de La Cavale Blanche, Brest
  - University Hospital Gabriel-Montpied, Clermond-Ferrand
  - University Hospital of Grenoble - Hôpital Sud, Échirolles
  - Le Mans Regional Hospital, Le Mans
  - Private Rheumatologist, Mantes-la-Jolie
  - University Hospital Lapeyronie, Montpellier
  - University Hospital Hotel-Dieu, Nantes
  - University Hospital Saint-Antoine, Paris
  - University Hospital La Pitié Salpétrière, Paris
  - University Hospital Cochin, Paris
  - University Hospital Sud, Rennes
  - University Hospital Purpan, Toulouse

REFERENCES:
- [Background] Maly RC, Frank JC, Marshall GN, DiMatteo MR, Reuben DB. Perceived efficacy in patient-physician interactions (PEPPI): validation of an instrument in older persons. J Am Geriatr Soc. 1998 Jul;46(7):889-94. doi: 10.1111/j.1532-5415.1998.tb02725.x. PMID 9670878
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Ann Rheum Dis. 2010 Sep;69(9):1580-8. doi: 10.1136/ard.2010.138461. PMID 20699241
- [Background] Gossec L, Dougados M, Rincheval N, Balanescu A, Boumpas DT, Canadelo S, Carmona L, Daures JP, de Wit M, Dijkmans BA, Englbrecht M, Gunendi Z, Heiberg T, Kirwan JR, Mola EM, Matucci-Cerinic M, Otsa K, Schett G, Sokka T, Wells GA, Aanerud GJ, Celano A, Dudkin A, Hernandez C, Koutsogianni K, Akca FN, Petre AM, Richards P, Scholte-Voshaar M, Von Krause G, Kvien TK. Elaboration of the preliminary Rheumatoid Arthritis Impact of Disease (RAID) score: a EULAR initiative. Ann Rheum Dis. 2009 Nov;68(11):1680-5. doi: 10.1136/ard.2008.100271. Epub 2008 Dec 3. PMID 19054825
- [Background] Pincus T, Bergman MJ, Yazici Y, Hines P, Raghupathi K, Maclean R. An index of only patient-reported outcome measures, routine assessment of patient index data 3 (RAPID3), in two abatacept clinical trials: similar results to disease activity score (DAS28) and other RAPID indices that include physician-reported measures. Rheumatology (Oxford). 2008 Mar;47(3):345-9. doi: 10.1093/rheumatology/kem364. Epub 2008 Jan 31. PMID 18238788
- [Background] Guillemin F, Braincon S, Pourel J. [Measurement of the functional capacity in rheumatoid polyarthritis: a French adaptation of the Health Assessment Questionnaire (HAQ)]. Rev Rhum Mal Osteoartic. 1991 Jun;58(6):459-65. French. PMID 1896787
- [Background] Smolen JS, Landewe R, Breedveld FC, Buch M, Burmester G, Dougados M, Emery P, Gaujoux-Viala C, Gossec L, Nam J, Ramiro S, Winthrop K, de Wit M, Aletaha D, Betteridge N, Bijlsma JW, Boers M, Buttgereit F, Combe B, Cutolo M, Damjanov N, Hazes JM, Kouloumas M, Kvien TK, Mariette X, Pavelka K, van Riel PL, Rubbert-Roth A, Scholte-Voshaar M, Scott DL, Sokka-Isler T, Wong JB, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs: 2013 update. Ann Rheum Dis. 2014 Mar;73(3):492-509. doi: 10.1136/annrheumdis-2013-204573. Epub 2013 Oct 25. PMID 24161836
- [Background] Bossert M, Prati C, Vidal C, Bongain S, Toussirot E, Wendling D. Evaluation of self-report questionnaires for assessing rheumatoid arthritis activity: a cross-sectional study of RAPID3 and RADAI5 and flare detection in 200 patients. Joint Bone Spine. 2012 Jan;79(1):57-62. doi: 10.1016/j.jbspin.2011.03.014. Epub 2011 May 6. PMID 21550283
- [Derived] Gossec L, Cantagrel A, Soubrier M, Berthelot JM, Joubert JM, Combe B, Czarlewski W, Wendling D, Dernis E, Grange L, Beauvais C, Perdriger A, Nataf H, Dougados M, Servy H. An e-health interactive self-assessment website (Sanoia(R)) in rheumatoid arthritis. A 12-month randomized controlled trial in 320 patients. Joint Bone Spine. 2018 Dec;85(6):709-714. doi: 10.1016/j.jbspin.2017.11.015. Epub 2017 Dec 12. PMID 29246532